CLINICAL TRIAL: NCT01124266
Title: Can Involvement of Endoscopy Nurse Participation Increase Adenoma Detection Rate During Screening Colonoscopy?:A Prospective Multicenter Randomized Trial
Brief Title: Endoscopy Nurse Participation in Adenoma Detection Rate During Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Soon Chun Hyang University (Other)
Collaborators: Kangbuk Samsung Hospital (Other); Hanyang University Guri Hospital (Other); Dankook University (Other); Incheon St.Mary's Hospital (Other); Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Chang Kyun Lee, MD, PhD, Soon Chung Hyang Universtiy, Cheonan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-15
Record Dates: First submitted 2010-05-14; First posted 2010-05-17 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2010-05

CONDITIONS: Polyp; Adenomatous Polyp; Colonoscopy
Keywords: polyp; adenoma; screening; colonoscopy; diagnosis
MeSH Terms: conditions — Polyps; Adenomatous Polyps; Adenoma; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- endoscopist only (Experimental)
  Interventions: Procedure: standard of care colonoscopy
- nurse participation (Experimental)
  Interventions: Procedure: standard of care colonoscopy

INTERVENTIONS:
Procedure: standard of care colonoscopy — Single inspection by endoscopist during colonoscopy
  Arms: endoscopist only
Procedure: standard of care colonoscopy — Dual inspection by both endoscopist and nurse during colonoscopy
  Arms: nurse participation

SUMMARY:
Colorectal cancer (CRC) is the second most common cancer and the fourth leading cause of cancer death in Korea. Colonoscopy with polypectomy decreases the incidence and mortality from colorectal cancer. However, significant lesions can be missed during colonoscopy. Recent retrospective studies have shown that fellow involvement as a second observer may increase adenoma detection rate in colonoscopy.

The aim of this prospective, multicenter, randomized study is to evaluate the impact when endoscopy nurse participate in adenoma detection during screening colonoscopy. The primary outcome measure is the adenoma detection rate (ADR).

ELIGIBILITY:
Inclusion Criteria:

* age over 50
* screening colonoscopy

Exclusion Criteria:

* History of colorectal surgery
* History of hereditary colorectal cancers or polyposis syndrome
* Gastrointestinal bleeding
* Inflammatory bowel diseases
* Inability to provide informed consent
* Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 844 (Actual)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
adenoma detection rate | 1 year

SECONDARY OUTCOMES:
subjects with at least one polyp | 1 year
Subjects with at least one adenoma | 1 year
total number of polyp | 1 year
total number of adenoma | 1 year
Subjects with at least one advanced adenoma or cancer | 1 year
total number of advanced adenoma or cancer | 1 year
polyp and adenoma detection rate according to the endoscopists or nurse experience | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chang Kyun Lee, MD, PhD, Principal Investigator — Soon Chun Hyang University
Locations (6):
- South Korea (6):
  - Dankook University Hospital, Cheonan
  - Soon Chun Hyang University Cheonan Hospital, Cheonan
  - Hanyang university Guri Hospital, Guri-si
  - The Catholic University Incheon St. Mary's Hospital, Incheon
  - Kangbuk Samsung Hospital, Seoul
  - Kyung Hee University Gangdong Hospital, Seoul

REFERENCES:
- [Background] Rogart JN, Siddiqui UD, Jamidar PA, Aslanian HR. Fellow involvement may increase adenoma detection rates during colonoscopy. Am J Gastroenterol. 2008 Nov;103(11):2841-6. doi: 10.1111/j.1572-0241.2008.02085.x. Epub 2008 Aug 27. PMID 18759826
- [Background] Peters SL, Hasan AG, Jacobson NB, Austin GL. Level of fellowship training increases adenoma detection rates. Clin Gastroenterol Hepatol. 2010 May;8(5):439-42. doi: 10.1016/j.cgh.2010.01.013. Epub 2010 Feb 1. PMID 20117245
- [Derived] Lee CK, Park DI, Lee SH, Hwangbo Y, Eun CS, Han DS, Cha JM, Lee BI, Shin JE. Participation by experienced endoscopy nurses increases the detection rate of colon polyps during a screening colonoscopy: a multicenter, prospective, randomized study. Gastrointest Endosc. 2011 Nov;74(5):1094-102. doi: 10.1016/j.gie.2011.06.033. Epub 2011 Sep 1. PMID 21889137